CLINICAL TRIAL: NCT06014099
Title: Research on the Application of Blood Collection Through Midline Catheters of Different Lengths
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhao Linfang, Assitant nursing director, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IV202308
Record Dates: First submitted 2023-03-13; First posted 2023-08-28 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Catheter Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Not possible because of the material and characteristics of the catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midline catheter (Experimental): The test group2 used MC for blood collection.
  Interventions: Behavioral: Midline catheter for blood collection
- Long peripheral venous catheters (Experimental): In the test 1 group, blood was collected using LPC.
  Interventions: Behavioral: Long peripheral venous catheters for blood collection
- short peripheral venous catheters (Other): In the control group,blood was collected using SPC.
  Interventions: Behavioral: SPCs for blood collection

INTERVENTIONS:
Behavioral: Long peripheral venous catheters for blood collection — used LPC for blood collection
  Arms: Long peripheral venous catheters
Behavioral: Midline catheter for blood collection — used MCs for blood collection
  Arms: Midline catheter
Behavioral: SPCs for blood collection — used SPCs for blood collection
  Arms: short peripheral venous catheters

SUMMARY:
Therefore, in this study, the investigators propose to use a randomized controlled prospective open study on inpatients with difficult blood collection, by comparing the effects of the application of two types of peripheral venous catheters for blood collection via LPC and MC, with a view to improving the success rate of blood collection in difficult peripheral venous blood collection, and providing a theoretical basis for the later application of long peripheral venous catheters and midline catheters; and providing a basis for optimizing the experience of venous blood collection by nurses.

DETAILED DESCRIPTION:
Using block randomization, patients were randomized in 1:1:1 blocks into experimental arm 1(Long peripheral venous catheter), experimental arm 2(midline catheter), and control (short peripheral venous catheter) with a block length of 6. Patients have a total of 27 blocks, import data into SPSS23, randomly group by SPSS, generate random numbers, and group according to the size of random numbers in each unit group, the largest in the group is assigned to the experimental group 1, the middle of the group is assigned to the experimental group 2, and the smallest in the group is assigned to the control group. The experimental group1 used the LPC for blood collection, the experimental group 2 used the MC for blood collection,and the control group used the Short PIVC for blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Meet the international diagnostic criteria for metabolic syndrome (such as ATP III criteria or domestic Diabetes Branch of Chinese Medical Association criteria).
* The estimated treatment time of intravenous infusion is 1-4 weeks, and the nature of the infusion drug meets the indications of LPCs and MCs.
* Blood samples should be collected more than 3 times during the hospital.

Exclusion Criteria:

* A history of radiotherapy, thrombosis, and trauma at the catheter site.
* Plan to discharge from the hospital with the tube.
* Vulnerable groups, including people with mental illness, cognitive impairment, critically ill patients, minors, pregnant women, illiterate, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-10-27 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of first blood collection | during catheter indwelling,an average of 2 weeks
  Number of successful initial venous blood collection cases as a percentage of the total number of cases in this group
Total success rate of blood collection | during catheter indwelling,an average of 2 weeks
  Number of patients with successful intravenous blood collection as a proportion of the number of cases in this group

SECONDARY OUTCOMES:
Catheter-related complication rate | during catheter indwelling,an average of 2 weeks
  The proportion of patients with complications as a proportion of the total number of cases
Number of days for catheters to linger | during catheter indwelling,an average of 2 weeks
  The number of days between catheter insertion and catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Linfang Zhao, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Linfang Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lima-Oliveira G, Lippi G, Salvagno GL, Picheth G, Guidi GC. Laboratory Diagnostics and Quality of Blood Collection. J Med Biochem. 2015 Jul;34(3):288-294. doi: 10.2478/jomb-2014-0043. Epub 2015 Jul 14. PMID 28356839
- [Background] HO Guidelines Approved by the Guidelines Review Committee[J]. 2015.
- [Background] Tsukuda Y, Funakoshi T, Nasuhara Y, Nagano Y, Shimizu C, Iwasaki N. Venipuncture Nerve Injuries in the Upper Extremity From More Than 1 Million Procedures. J Patient Saf. 2019 Dec;15(4):299-301. doi: 10.1097/PTS.0000000000000264. PMID 27314202
- [Background] Jeong Y, Park H, Jung MJ, Kim MS, Byun S, Choi Y. Comparisons of laboratory results between two blood samplings: Venipuncture versus peripheral venous catheter-A systematic review with meta-analysis. J Clin Nurs. 2019 Oct;28(19-20):3416-3429. doi: 10.1111/jocn.14918. Epub 2019 Jun 10. PMID 31112315
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Background] Wicker S, Stirn AV, Rabenau HF, von Gierke L, Wutzler S, Stephan C. Needlestick injuries: causes, preventability and psychological impact. Infection. 2014 Jun;42(3):549-52. doi: 10.1007/s15010-014-0598-0. Epub 2014 Feb 14. PMID 24526576
- [Background] Zhang Y, Zhang S, Chen J, Zhao R. Blood sampling from peripherally inserted central catheter is effective and safe for patients with head and neck cancers. J Vasc Access. 2021 May;22(3):424-431. doi: 10.1177/1129729820943458. Epub 2020 Aug 3. PMID 32741243